CLINICAL TRIAL: NCT00868114
Title: A Phase II Study of Apoptosis Induction Through Direct Tumor Injection of TNFerade(TM)or Radiation Alone Followed by KLH-Pulsed Autologous Dendritic Cells in Patients With Unresectable Pancreatic Cancer
Brief Title: Direct Tumor Injection KLH-Pulsed Dendritic Cells in Unresectable Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Leo W. Jenkins Cancer Center (Other)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LJCC 09-01; RCA115018B
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Inoperable pancreatic cancer; Dendritic Cell Vaccine; Locally advanced or low volume metatstatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 3 weekly injections of intratumoral TNFerade plus radiation and 3 weekly intratumoral injections of dendritic cell vaccine
  Interventions: Biological: KLH-pulsed autologous dendritic cell vaccine
- 2 (Experimental): Radiation Only with 3 weekly intratumoral injections of dendritic cell vaccine
  Interventions: Biological: KLH-pulsed autologous dendritic cell vaccine

INTERVENTIONS:
Biological: KLH-pulsed autologous dendritic cell vaccine — 5 X10e7 KLH-pulsed autologous dendritic cell vaccine once weekly times three weeks

SUMMARY:
This research study uses radiation or a gene therapy agent, TNFerade in addition to a dendritic cell vaccine in patients with locally advanced or low volume metastatic pancreatic cancer. The use of TNFerade or radiation serves to generate cell death stimulating the immune response. The dendritic cell vaccine may direct a distant and lasting effective anti-tumor immune response to achieve a local and systemic clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven, unresectable pancreatic cancer with an intact primary tumor that is accessible to direct intratumoral injection
* Low volume metastatic disease defined as 1) radiographically occult disease discovered at the time of anticipated resection or 2) no more than 4 radiographically detected metastasis none of which are greater than 2 cm in greatest dimension
* Good overall health with a Karnofsky performance status of 70% or greater
* No evidence or history of an autoimmune dysfunction
* Life expectancy > 3 months
* Agreement to initiate and complete standard treatment (chemotherapy ± radiation) for pancreatic cancer at the completion of the study
* Age equal to or greater than 18 years
* No prior or concurrent chemotherapy
* No previous or concurrent immunotherapy for pancreatic cancer
* Liver enzymes ≤ 3 times upper limit of normal:
* Tbili ≤ 3.9 (biliary stents are allowed)
* AST ≤ 177
* ALT ≤ 198
* Alk phos ≤ 378
* Adequate pretreatment organ function:

  * Creatinine no greater than 1.5mg/dL
  * Total calcium no greater than 11.0mg/dL
  * PT no greater then 14 seconds
  * PTT no greater then 40 seconds
* Ability to give informed consent
* Adequate baseline hematopoietic function:

  * Total white blood cell count equal to or greater than 3,000/mm3;
  * Absolute granulocyte count greater than 1,500/mm3;
  * Absolute lymphocyte count greater than 500/mm3;
  * Platelet count equal to or greater than 100,000/mm3.

Exclusion Criteria:

* Prior history of XRT to primary pancreatic tumor
* Patients with tumors that are not accessible to direct access cannot be included in the study, nor will patients with poor overall health as determined by standard laboratory data and performance scales
* Prior or concurrent chemotherapy
* Prior history (within last four weeks) of antineoplastic therapy or irradiation
* Prior treatment with anti-tumor vaccines not allowed
* Patients with a history of autoimmune diseases such as SLE, rheumatoid arthritis or myasthenia gravis
* A history of HIV infection, AIDS or other immunosuppressive disease state
* Patients requiring regular corticosteroids within the past year are ineligible. There must be no use of corticosteroids in the fours weeks preceding entry into the study
* Active bacterial, fungal or viral infection
* Active bleeding (hemoptysis, melena, etc)
* Women who are currently pregnant or actively breast feeding. Women of childbearing potential must have a negative serum pregnancy test and must use effective contraception during trial participation
* Uncontrolled or unstable medical conditions, including angina, bronchospasm, hypertension, hyperglycemia, hypercalcemia and cardiac arrhythmia
* Any medical or psychiatric illness which in the opinion of the principal investigator might compromise a patient's ability to tolerate or complete treatment
* Patients requiring anticoagulation are ineligible
* Refusal to receive standard treatment (chemotherapy ± radiation) after the completion of the protocol
* Evidence of DVT or prior history of DVT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-07; Primary Completion 2013-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Patients will be followed until death

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel E Zervos, MD, Principal Investigator — East Carolina University - Leo W. Jenkins Cancer Center
Locations (1):
- East Carolina University - Leo W. Jenkins Cancer Center, Greenville, North Carolina, United States